CLINICAL TRIAL: NCT06559592
Title: Internal Unicompartmental Arthroplasty After Tibial Valgization Osteotomy
Acronym: ArOs
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: ArOs (29BRC21.0209)
Record Dates: First submitted 2022-08-04; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2022-05

CONDITIONS: Knee Arthritis
Keywords: orthopedic surgery; unicompartmental knee arthroplasty; high tibial osteotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This retrospective, monocentric study is about outcomes concerning patients who benefit from medial unicompartmental knee arthroplasty after previous high tibial osteotomy. This previous high tibial osteotomy was performed because of genu varum.

Clinical, funtionnal and radiological outcomes were examined.

ELIGIBILITY:
Inclusion Criteria:

* operated between January 2005 and June 2019
* HTO followed by implantation of medial UKA (Oxford Partial Knee, Zimmer Biomet, Bridgend, UK) in the same knee
* medial knee osteoarthritis with healthy lateral compartment
* patellofemoral pain
* coronal plane deformity of less than 15°

Exclusion Criteria:

* death
* lost to follow-up
* medial UKA implant other than the Oxford Partial Knee

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients aged of at least18 years old, who benefit from medial unicompartmental knee arthroplasty after previous high tibial osteotomy. The high tibial osteotomy was made because of genu varum.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-11-02 (Actual)

PRIMARY OUTCOMES:
Give the functional results using the Oxford score, for patients who underwent this procedure. | from 4 to 185 months
  Oxford Knee Scale (OKS) score results after a mean follow-up of 79 months after unicompartmental internal arthroplasty, and a mean follow-up of 185 months after tibial valgization osteotomy

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending five years maximum following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. requestors will be required to sign and complete a data access agreement